CLINICAL TRIAL: NCT06717373
Title: Point-of-Care Echocardiography in Patients with Known or Suspected Aortic Stenosis
Acronym: POC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caption Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CH_AutoAS_2024
Record Dates: First submitted 2024-07-19; First posted 2024-12-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Patients with an Indication for an Echocardiographic Examination with Suspicion of Valcular Heart Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, un-blinded study in patients scheduled for a standard echocardiographic examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Other): There is no investigational device being used. Devices to be used are Vscan Air and Venue Ultrasound systems
  Interventions: Device: AutoAS

INTERVENTIONS:
Device: AutoAS — AutoAS is an artificial intelligence algorithm that will be tested retrospectively on the images acquired as part of the study

SUMMARY:
This is a prospective clinical trial intended to capture echocardiographic images in patients clinically indicated for an echocardiographic examination using an additional Point of Care Ultrasound device . The images collected will be used to test and possibly validation an AI base Aortic Valve Stenosis algorithm

DETAILED DESCRIPTION:
This is a non-randomized, un-blinded single-arm study in patients scheduled for a standard echocardiographic examination. Participants will be scanned by a sonographer (Study Exam) and 6 standard views will be obtained using both the ultrasound systems: PLAX, PSAX-AV, AP4, AP2, AP3 and AP5 .

The patient will undergo their scheduled echocardiographic examination either before or after the study examinations.

The findings from the clinically indicated echocardiographic examination will be used as a gold standard for the presence/absence and severity of aortic stenosis.

The first 45 patients, 15 with mild, 15 with moderate and 15 with severe AS, will be used for testing and possible fine-tuning the AutoAS algorithm for each Study Device, and the remaining up to 155 patients for each Study Device will be used for clinical validation of the algorithm. Because these first 45 patients will only be used for possible fine-tuning the AutoAS algorithm, they will be excluded from endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an echocardiographic examination
* Patients ≥18 years old
* Patient with known or suspected valve disease based on medical history

Exclusion Criteria:

* Patients with artificial aortic valves
* Unable to lie flat for study
* Patients experiencing a known or suspected acute cardiac event
* Patients unwilling or unable to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | At the time of the examination
  The primary endpoints are the sensitivity and specificity of the Caption AutoAS algorithm for the absence (none/mild AS) or presence (moderate/severe AS) of AS relative to that indicated in the echocardiographic examination.

SECONDARY OUTCOMES:
Subgroup analysis of outcome 1 | At the time of the examination
  Subgroup Analyses: Sensitivity and specificity will be calculated for the following sub-groups. BMI group (< 25, ≥ 25-30, ≥ 30), sex, and age (<65, ≥65)

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Narang, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No